CLINICAL TRIAL: NCT04631237
Title: Developing a Down Syndrome Health Instrument
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Stephanie Santoro, Assistant Professor of Pediatrics, Clinical Geneticist, Massachusetts General Hospital
Other Study IDs: 2020P000213
Record Dates: First submitted 2020-10-22; First posted 2020-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Down Syndrome; Health, Subjective
Keywords: health status
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Focus Groups: N=52
  Interventions: Other: Observational, no intervention
- Cognitive Interviews: N=24
  Interventions: Other: Observational, no intervention
- Survey: N=542
  Interventions: Other: Observational, no intervention

INTERVENTIONS:
Other: Observational, no intervention — No intervention involved

SUMMARY:
Although over 200,000 individuals with DS live in the United States, studies to date have focused on outcomes apart from health. The foundation for this proposal is based on the need to accurately measure health of all individuals - specifically, with DS - and the dearth of available tools for this population. Creating such an instrument will provide a barometer of the current state of health for DS and hold use in future research. In this project, I propose to create an instrument that directly assesses health in DS - the Down syndrome Health Instrument (DHI). More specifically, the aims of this proposal are: 1. To conduct focus groups among caregivers, individuals with DS, panels of experts on DS and primary care physicians, and cognitive interviews to refine a conceptual model of health for DS and create an item pool, 2. To administer the DHI and establish internal validity, reliability, and external validity of the DHI for use in clinical research, and 3. To test the usability of the DHI in two pilot settings: research and clinical. This instrument will measure patient-reported health in DS for the first time and allow measurement of health as an outcome which is not currently possible in this population. This can identify gaps in care, then direct and optimize interventions that will improve care.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of an individual with DS (individual with DS age: <22 years)
* Caregiver age: ≥18 years
* Fluent in written and spoken English
* Able to read and provide informed consent

Exclusion Criteria:

* Physical or mental condition of caregiver that would prohibit self-administration of questionnaire
* Mosaic Down syndrome: based on medical record review. If caregiver is uncertain or mosaicism is unknown, we will request additional records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary caregivers and individuals with DS
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Survey results, cognitive interviews, and validation | Within 12 months of completion of analysis of surveys
  Local and national survey results, cognitive interviews and validation of DHI

SECONDARY OUTCOMES:
Focus group results and conceptual model | Within 12 months of completion of focus groups
  Descriptive focus group results regarding health views. Outline of the preliminary conceptual model

CONTACTS AND LOCATIONS:
Overall Officials: STEPHANIE L SANTORO, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santoro SL, Peters MLB. K Awards: The Journey of a Thousand Steps. Ann Intern Med. 2021 Dec;174(12):1735-1737. doi: 10.7326/M21-2692. Epub 2021 Nov 16. No abstract available. PMID 34781710
- [Result] Santoro SL, Donelan K, Constantine M. Proxy-report in individuals with intellectual disability: A scoping review. J Appl Res Intellect Disabil. 2022 Sep;35(5):1088-1108. doi: 10.1111/jar.13013. Epub 2022 Jun 8. PMID 35676858
- [Result] Santoro SL, Cabrera MJ, Haugen K, Krell K, Merker VL. Indicators of health in Down syndrome: A virtual focus group study with patients and their parents. J Appl Res Intellect Disabil. 2023 Mar;36(2):354-365. doi: 10.1111/jar.13065. Epub 2023 Jan 9. PMID 36624557
- [Result] Santoro SL, Cabrera MJ, Co JPT, Constantine M, Haugen K, Krell K, Skotko BG, Winickoff JP, Donelan K. Health in Down syndrome: creating a conceptual model. J Intellect Disabil Res. 2023 Apr;67(4):323-351. doi: 10.1111/jir.13007. Epub 2023 Jan 17. PMID 36650105
- [Result] Santoro SL, Haugen K, Donelan K, Skotko BG. Global health measures from a National Down Syndrome Registry. Am J Med Genet A. 2023 Aug;191(8):2092-2099. doi: 10.1002/ajmg.a.63243. Epub 2023 May 14. PMID 37183579
- [Result] Shaffer M, Co JPT, Donelan K, Skotko BG, Torres A, Winickoff JP, Santoro SL. Successful (and Unsuccessful) Recruitment Approaches and Participant Loss in a Down Syndrome Survey. Am J Intellect Dev Disabil. 2025 Mar 1;130(2):131-145. doi: 10.1352/1944-7558-130.2.131. PMID 39999870
- [Result] Witt M, Shaffer M, Torres A, Santoro SL. Research Letter: Recruiting a Diverse Cohort in Genetics Research-Reflecting on Demographic Representation in a Down Syndrome Survey. Am J Med Genet A. 2025 Oct;197(10):e64111. doi: 10.1002/ajmg.a.64111. Epub 2025 May 20. No abstract available. PMID 40391503
- [Result] Witt M, Palumbo M, Santoro SL. Bothersome and Impactful Health Conditions in Children and Adolescents with Down Syndrome. J Pediatr. 2025 Dec;287:114748. doi: 10.1016/j.jpeds.2025.114748. Epub 2025 Jul 23. PMID 40712746
- [Result] Witt M, Krell K, Santoro SL. Caregiver Interviews Regarding Health in Down Syndrome. Am J Med Genet A. 2026 Feb;200(2):300-307. doi: 10.1002/ajmg.a.64253. Epub 2025 Sep 12. PMID 40937636
- [Result] Santoro SL, Nichols D, Witt M, Oreskovic NM. Daily Activities, Exercise and Endurance in Down Syndrome. Am J Med Genet A. 2025 Oct 16:e64283. doi: 10.1002/ajmg.a.64283. Online ahead of print. PMID 41098034
- [Derived] Krell K, Witt M, Santoro SL. Caregivers' Perspectives on Medical Management and Its Helpfulness in Down Syndrome. Am J Med Genet A. 2025 Nov 27:e70006. doi: 10.1002/ajmga.70006. Online ahead of print. PMID 41306073
- [Derived] Santoro SL, Campbell A, Cabrera M, Co JPT, Donelan K, Haugen K, Krell K, Shaffer M, Skotko BG, Winickoff JP, Witt M, Constantine M. Development and Validation of a Health Measure for Down Syndrome. J Pediatr. 2025 Nov 4;289:114888. doi: 10.1016/j.jpeds.2025.114888. Online ahead of print. PMID 41192789

DOCUMENTS (2):
  • Informed Consent Form: Study information sheet (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT04631237/ICF_000.pdf
  • Informed Consent Form: Online consent form (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04631237/ICF_001.pdf